CLINICAL TRIAL: NCT04974463
Title: Using Genomics and Gut Microbiome Data to Predict Postoperative Opioid Use in Patients Undergoing Lower Extremity Joint Replacement
Brief Title: Predicting Chronic Opioid Use Following Lower Extremity Joint Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rodney Gabriel, Associate Professor, University of California, San Diego
Other Study IDs: 210132
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Joint Pain; Chronic Pain; Opioid Use
MeSH Terms: conditions — Arthralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — we will receive pharmacogenomic (blood), microbiome, and microsomal exosome samples from subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persistent Opioid Use at 3 months: Patients who continue to use opioids about 3 months after their joint replacement surgery
- No Persistent Opioid Use at 3 months: Patients who do not use opioids after about 3 months following joint replacement surgery

SUMMARY:
Personalized medicine is a concept in which medical care is individualized to a patient based on their unique characteristics, including comorbidities, demographics, genetics, and microbiome. After major surgery, some patients are at increased risk of opioid dependence. By identifying unique genetic and microbiome markers, clinicians may potentially identify individual risk factors for opioid dependence. By identifying these high risk patients early-on, personalized interventions may be applied to these patients in order to reduce the incidence of opioid-dependence.

DETAILED DESCRIPTION:
The primary objective of this study is to identify associations with genetic variants, gut microbiome, and metabolomics (i.e. exosome profiling) with postoperative opioid use in surgical patients. Patients will be recruited preoperatively who underwent lower extremity joint replacement. The following tests will be performed: 1) genome-wide single nucleotide polymorphisms and structural variation, with a particular focus on the following genes: COMT, BDNF, SCN11a, OPRM1, ACBC1, CYPD26, CYP34A, ANKK1, OPRD1, OPRK1,NGFB, UGT2B7, FFAR2, FFAR3, GABRG2, SLCO1B1, DRD4; 2) longitudinal gut microbiome sampling; and 3) exosome profiling - blood will be collecting for RNAseq and plasma for metabolomics and extracellular vesicle characterization with ultimate impact on in vitro cell function. These genes were selected because they have been shown to be associated with opioid use, opioid metabolism, and pain. Furthermore, subjects will fill out surveys preoperatively, including: pain catastrophizing scale, brief pain inventory, PROMIS-29, and fibromyalgia survey criteria. Other data collected will include body mass index, age, sex, comorbidities, lifestyle habits, and medication use.

The hypothesis is that there will be clinically significant associations with patient genetics, microbiome, exosome profiles with their postoperative opioid use. Such findings will help personalize pain interventions for high-risk patients undergoing knee or hip arthroplasty in order to help improve postoperative pain control and reduce incidence of chronic opioid use.

Specific Aim #1. To validate and identify pharmacogenomic associations with acute postoperative opioid use (during the first 48 postoperative hours) and chronic opioid use (at >3-4 months after surgery) in patients who underwent lower extremity joint replacement.

Specific Aim #2. To identify gut microbiome and metabolomics associations with acute postoperative opioid use (during the first 48 postoperative hours) and chronic opioid use (at >3-4 months after surgery) in patients underwent lower extremity joint replacement.

Specific Aim #3. To identify blood RNAseq patterns, plasma metabolic markers, extracellular vesicles, and impact of plasma on in vitro cell metabolism associated with acute postoperative opioid use (during the first 48 postoperative hours) and chronic opioid use (at >3-4 months after surgery) in patients underwent lower extremity joint replacement.

Machine learning approaches will be used to combine all data to improve prediction of the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing unilateral knee or hip arthroplasty

Exclusion Criteria:

* refusal to consent
* lack of independent decision-making capacity
* inability to communicate effectively with research personnel
* if patient received antibiotics within the last 3 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing lower extremity joint replacement (i.e. total knee arthroplasty, total hip arthroplasty, hemiarthroplasty, unicompartmental knee replacement)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
3-month persistent opioid use | 3 months
  continual opioid use 3 months after surgery
3-month persistent post-surgical pain | 3 months
  continual pain at surgical site at 3 months

SECONDARY OUTCOMES:
Acute postoperative opioid use | 48 hours
  opioid use during the first 48 hours after surgery
Acute postoperative pain | 48 hours
  pain scores during the first 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided